CLINICAL TRIAL: NCT04536467
Title: Prevention of Chemotherapy-Induced Ovarian Failure With Goserelin in Premenopausal Lymphoma Patients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, ALshaimaa Ibrahim Rabie, clinical pharmacy department, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA 00015574
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Goserelin; Drug Therapy; Antineoplastic Combined Chemotherapy Protocols

STUDY DESIGN:
Intervention Model Description: Arm 1: Goserelin plus standard chemotherapy Arm 2 (control Arm): Standard chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goserelin arm (Other): 3.6 mg subcutaneous injection in the abdominal wall every 4 weeks (28 ± 3 days) plus standard chemotherapy at start of regimen for 3 months
  Interventions: Drug: Goserelin
- control Arm (Other): Standard chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Goserelin — chemotherapy+goserelin
  Other Names: zoladex
  Arms: Goserelin arm
Drug: Chemotherapy — standard chemotherapy
  Other Names: chemotherapy protocols
  Arms: control Arm

SUMMARY:
To Prevent Chemotherapy Induced Ovarian Failure with the gonadotropin-releasing hormone Agonist Goserelin in Young female Lymphoma Cancer patients Receiving Chemotherapy

DETAILED DESCRIPTION:
Design:

Study will be prospective interventional simple randomized control parallel open label Arms and Interventions Arm 1: Goserelin plus standard chemotherapy Goserelin will be given as a 3.6 mg subcutaneous injection in the abdominal wall every 4 weeks (28 ± 3 days) plus standard chemotherapy at start of regimen for 3 months (26) Arm 2 (control Arm): Standard chemotherapy Patients will take only standard chemotherapy for 3 months Setting: oncology department Beni Suef university hospital Sample size: 80 patients (based on the results from the literature and to ensure a power of 80% and a type I error probability of 5%. we calculate Effect size Primary Outcome Measures

Evaluating ovarian function by: at the start of treatment and after 3 cycles chemotherapy treatment and at end of 6 cycles chemotherapy through:

* FSH level (follicle-stimulating hormone (FSH))
* Estradiol level
* AMH level follow up time time frame 1 year follow up after chemotherapy

Secondary Outcome Measures:

* Overall All Response determined by tumor assessments from radiological tests including one of the following (computed tomography scan, Magnetic resonance imaging Positron-emission tomography or physical examinations according RECIL 2017 criteria.
* Adverse events (Sweating, Hot flushes, vaginal bleeding, vaginal dryness. Headaches)

ELIGIBILITY:
Inclusion Criteria:

Female lymphoma patients will be included in the study if they meet the following criteria:

1. Confirmed lymphoma cancer radiological and pathological or by clinical evaluation receiving chemotherapy treatment
2. Normal FSH-level , estradiol level (FSH levels less than 10IU/L at the time of random assignment)
3. Female Age between 17- 40 years
4. Written informed consent

Exclusion criteria:

The patients will be excluded from the study if they have the following criteria:

1. Known hypersensitivity reaction to the investigational compounds or incorporated substances
2. Primary ovarian dysfunction, previous history of amenorrhea >3 months
3. Age > 40
4. Pregnant or lactating patients, prior use of hormonal contraceptives has to be discontinued before first Goserelin injection
5. patients who are unlikely to comply with trial requirements (eg, confusion, psychological or mood disturbances ,alcoholism, Vaginitis, vaginal bleeding, cardiac arrhythmia)

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — woman age 17-40 years
Enrollment: 80 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
prevention premature ovarian failure | 6 month from start of chemotherapy
  Evaluating ovarian function by FSH,E2 levels

SECONDARY OUTCOMES:
overall response in lymphoma patients | 6 month
  Overall response rate determined by tumor assessments from radiological tests including one of the following (computed tomography scan, Magnetic resonance imaging Positron-emission tomography or physical examinations , ( RECIL 2017) The overall response evaluation criteria in lymphoma, criteria categorized patients stable disease,progressive disease ,minor response,partial response,complete response at end of 6 months.
ADVERSE EFFECTS | 6 MONTH
  Adverse events (Sweating, Hot flushes, vaginal bleeding, vaginal dryness. Headaches)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdullah Elberry Elberry, MD, Study Director — Assistant Professor of Clinical Pharmacology, Beni-Suef University; Raghda Roshdy Sayed Hussein, MD, Study Director — Lecturer of Clinical pharmacy, Beni-Suef University; ahmed hassan shaaban, Study Director — Lecturer of Clinical Oncology, Beni-Suef University
Locations (1):
- Beni Suef university, Al Fayyum, Mesala, Egypt

IPD SHARING:
Plan to Share IPD: No